CLINICAL TRIAL: NCT04061395
Title: Guselkumab for Hidradenitis Suppurativa, a Mode of Action Study. The HiGUS-trial
Brief Title: Guselkumab for Hidradenitis Suppurativa, a Mode of Action Study.
Acronym: HiGUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CNTO1959HDS2002
Record Dates: First submitted 2019-08-09; First posted 2019-08-19 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Guselkumab (Experimental): Guselkumab 200 mg Q4W; subcutaneous injections; duration of 16 weeks.
  Interventions: Biological: Guselkumab

INTERVENTIONS:
Biological: Guselkumab — See study arm description.
  Other Names: Tremfya

SUMMARY:
This is a multicenter open-label mode of action study. Twenty patients with moderate to severe hidradenitis suppurativa will be treated with guselkumab 200 mg Q4W subcutaneously. Main objectie is to investigate changes in inflammatory pathways induced by IL-23p19 blockade with guselkumab, in HS lesional skin.

The total duration of the treatment period per subject is 16 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* moderate to severe HS
* treatment history of at least one systemic anti-inﬂammatory / immunosuppressive agent;
* HS diagnosis of at least 1 year;
* minimum of two anatomical locations with HS lesions
* minimum of 4 active abscesses and/or inflammatory nodules (AN).

Key Exclusion Criteria:

* contra-indication for guselkumab;
* previous use of guselkumab;
* use of treatment with biologics or any immunosuppressives for HS in the last 3 months prior to randomization;
* presence of other uncontrolled major disease;
* pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in inflammatory pathways induced by IL-23p19 blockade with guselkumab. | Week 0 and 16
  Pangenomic gene expression profiling at week 0 and week 16 will be performed on skin biopsies to investigate changes in levels of cytokines in the skin.

SECONDARY OUTCOMES:
Clinical efficacy - Inflammatory lesion count and Hidradenitis Suppurativa Clinical Response (HiSCR) | Week 0, 4, 12, 16.
  All inflammatory lesions on all affected body areas will be counted. Additionally, the HiSCR will be calculated from these counted lesions.
Clinical efficacy - International Hidradenitis Suppurativa Severity Score System (IHS4). | Week 0, 4, 12, 16.
  The IHS4 score will be calculated by multiplying the number of nodules by 1, the number of abscesses by 2 and the number of draining fistulas by 4 and adding up these three outcomes into a total score.
Patient reported outcomes - Patient Global Assessment | Every four weeks
  Patient will be asked to assess his or her skin disease activity with in 5 categories.
Patient reported outcomes - Itch Numeric Rating Scale | Week 0, 4, 8, 12 and 16
  Patient will be asked to score his or her itch on numeric rating scale from 0 (no itch) to 10 (worst possible itch).
Patient reported outcomes - Pain Numeric Rating Scale | Week 0, 4, 8, 12 and 16
  Patient will be asked to score his or her pain on numeric rating scale from 0 (no pain) to 10 (worst possible pain).
Patient reported outcomes - Patient treatment satisfaction score | Week 0 and 16
  Patient will be asked to score his or her satisfaction about the treatment at baseline and at week 16 on a numeric rating scale from 0 (completely unsatisfied) to 10 (completely satisfied).
Patient reported outcomes - Dermatology Life Quality Index | Week 0, 4, 8, 12 and 16
  A survey containing 10 questions regarding multiple aspects of the quality of life. Each question has 4 answer possibilities: 'not at all', 'a little', 'a lot' and 'very much'. These answers correspond with 0,1,2 or 3 points respectively. The total score can range from 0 to 30 points.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Erasmus MC, University Medical Center Rotterdam, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen